CLINICAL TRIAL: NCT03423706
Title: Clinical Studies of New Model Haploidentical Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART
Record Dates: First submitted 2018-01-16; First posted 2018-02-06 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-01

CONDITIONS: CD19-chimeric Antigen Receptor T Cells; Relapsed and/or Refractory Acute Lymphoblastic Leukemia; the Haploidentical Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- new model of haplo-HSCT (Experimental): use the new model of haplo-HSCT to treat the r/r B-ALL patients matching the inclusion criterion
  Interventions: Procedure: the new model of haplo-HSCT for r/r B-ALL

INTERVENTIONS:
Procedure: the new model of haplo-HSCT for r/r B-ALL — take advantage of high-dose CTX、CD19-CART、donor CD34+HSC and Tregs to create a new model of haplo-HSCT for the patients in r/r B-ALL,to improve the quality of HSCT.

SUMMARY:
Building a new haploid transplanted model with high-dose CTX、CD19-CART,donor CD34+ hematopoietic stem cell and Tregs,to prevent graft-versus-host disease(GVHD),reduce the infection,promote the rate of immune reconstruction，seperate graft versus leukemia（GVL）and GVHD，then to reduce the relapse rate after hematopoietic stem cell transplantation（HSCT）for relapsed and/or refractory B cell acute lymphoblastic leukemia（r/r-B-ALL）.

DETAILED DESCRIPTION:
compare the new haplo-HSCT model with the traditional haplo-HSCT in DFS、OS、RFS、CR and the degree of GVHD.etc.for the r/r B-ALL patients.

ELIGIBILITY:
Inclusion Criteria:

1. the r/r B-ALL patients
2. have the healthy allo-HSCT donor
3. voluntary and signed the treatment protocol

Exclusion Criteria:

1. not match the inclusion criteria
2. important organ is dysfunction, such as heart and/or renal dysfunction,liver failure
3. Pregnancy or breast-feeding women
4. has virus infection,such as HIV,hepatitis virus,and can not be cleared with anti-virus treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-05-07 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
disease free survival at six months | six months
  the disease free survival of the new model haplo-HSCT will be assessed at 6 months.
acute graft-versus-host disease | three months
  we will examine the treatment-related acute GVHD at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: jin zhou, doctor, Study Chair — First affliliated hospital of Harbin medical university
Locations (1):
- First affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China